CLINICAL TRIAL: NCT02902601
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability, and Pharmacodynamics of JNJ-54175446 in Subjects With Major Depressive Disorder
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacodynamics of JNJ-54175446 in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108204; 54175446MDD1001 (Other: Janssen Research & Development, LLC); 2016-001929-14 (EudraCT Number)
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — JNJ-54175446

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Group A: JNJ-54175446 (Experimental): Participants will receive a loading dose of JNJ-54175446, 600 milligram (mg) on Day 1 followed by JNJ-54175446, 150 mg once daily until Day 10.
  Interventions: Drug: JNJ-54175446, 600 mg; Drug: JNJ-54175446, 150 mg
- Group B: Placebo + JNJ-54175446 (Experimental): Participants will receive placebo on Days 1 to 3 followed by a loading dose of JNJ-54175446, 600 mg on Day 4 followed by JNJ-54175446, 150 mg once daily until Day 10.
  Interventions: Drug: JNJ-54175446, 600 mg; Drug: JNJ-54175446, 150 mg; Other: Placebo
- Group C: Placebo (Placebo Comparator): Participants will receive placebo from Day 1 until Day 10.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JNJ-54175446, 600 mg — Participants will receive JNJ-54175446, 600 mg as an oral suspension.
  Arms: Group A: JNJ-54175446; Group B: Placebo + JNJ-54175446
Drug: JNJ-54175446, 150 mg — Participants will receive JNJ-54175446, 150 mg as an oral suspension.
  Arms: Group A: JNJ-54175446; Group B: Placebo + JNJ-54175446
Other: Placebo — Matching placebo to JNJ-54175446
  Arms: Group B: Placebo + JNJ-54175446; Group C: Placebo

SUMMARY:
The primary purpose of this study is to investigate the safety and tolerability of JNJ 54175446 in participants with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) must be between 18 and 32 kilogram per square meter (kg/m^2) inclusive
* Related to symptoms of depression: Participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV or V diagnostic criteria for Major Depressive Disorder [MDD] (International Classification of Diseases (ICD)-code F32.x and F33.x), without psychotic features, as confirmed by the MINI 6.0; participant must have an IDS-C30 total score greater than or equal to (>=) 30 using the semi-structured interview guide for the IDS-C30
* Participant is, during this episode of depression, treatment naïve OR treated with at most one Selective serotonin reuptake inhibitor (SSRI) over a minimum of 6 weeks and a maximum of 6 months, and subject is being treated at an adequate dose, showing a partial response at enrolment
* A woman of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test upon admission
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Has a primary DSM-IV or V diagnosis of general anxiety disorder (GAD), panic disorder, obsessive compulsive disorder, posttraumatic stress disorder, anorexia nervosa, or bulimia nervosa. Participants with comorbid GAD, social anxiety disorder, or panic disorder for whom MDD is considered the primary diagnosis are not excluded
* Has a length of current major depressive episode greater than (>) 24 months despite adequate treatment
* Has failed more than 2 treatments with a different pharmacological mode of action despite an adequate dose and duration during a previous, or the current depressive episode
* Participant has a history of substance use disorder according to DSM-V criteria, except nicotine or caffeine, within 6 months before Screening. However, participants who have completed a treatment for (alcohol) addiction more than 8 weeks prior to first dose administration and are under continuous control of the study center, may be included if the risk to fall back is considered minimal and no significant abnormalities are shown in clinical laboratory or other predose safety assessments
* Obstructive sleep apnea/hypopnea (apnea/hypopnea index >10) or restless legs syndrome (periodic leg movements with arousal index >15) as assessed on the first or second polysomnography (PSG) recording during screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 17

SECONDARY OUTCOMES:
Effect of JNJ-54175446 Versus Placebo on Total Sleep Deprivation (TSD)-Induced Changes in Depressive Symptoms by HDRS17/IDS-C30 Rating Scale | Baseline, Day 4 and 10: 2 to 8 hours post dose, Day 17
  Hamilton Depression Rating Scale 17 (HDRS17) contains 17 items pertaining to symptoms of depression experienced over the past week. Score range is from 0 to 52. The Inventory of Depressive Symptomatology- Clinician rated-30 (IDS-C30) is a standardized 30 item, clinician rated, scale to assess the severity of a participant's depressive symptoms. The scores range from a minimum of 0 to a maximum score of 84. The higher the score the more severe the symptoms of depression.
Effect of JNJ-54175446 Versus Placebo on Total Sleep Deprivation (TSD)-Induced Changes in Depressive Symptoms by QIDS-SR16/QIDS-SR10 Rating Scale | Baseline, Day 3 and 10: 2 to 8 hours post dose, Day 17
  The QIDS-SR16 (1 week recall period) is a participant reported measure designed to assess the severity of depressive symptoms. The total score ranges from 0 to 27 (none 1-5, mild 6-10, moderate 11-15, severe 16-20 and very severe 21-27). QIDS-SR10 is a version of the QIDS-SR16 with a shorter, 2-hour recall period and 10-item measure. Scoring for each domain will be the same as for the QIDS-SR16.
Effect of JNJ-54175446 Versus Placebo on TSD-Induced Changes in Biomarker Profiles (interleukin [IL]-1 beta, cortisol) | Day 1 and 4: Predose, 2, 8 hours postdose, Day 10: Predose
Effect of JNJ-54175446 Versus Placebo on Latency to Persistent Sleep (LPS) | Baseline, Day 2 to 3 and Day 4 to 5
  Latency to persistent sleep is defined as the length of time from full wakefulness to the first sleep stage.
Effect of JNJ-54175446 Versus Placebo on Total Sleep Time (TST) | Baseline, Day 2 to 3 and Day 4 to 5
  All of the minutes of Stages 1, 2, 3/4 Non Rapid Eye-Movement (NREM) and Rapid-Eye-Movement (REM) sleep, as measured by Polysomnography, are summed to determine the Total Sleep Time.
Effect of JNJ-54175446 Versus Placebo on Wake After Sleep Onset (WASO) | Baseline, Day 2 to 3 and Day 4 to 5
  The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Effect of JNJ-54175446 Versus Placebo on Sleep Efficiency (SE) | Baseline, Day 2 to 3 and Day 4 to 5
  The total sleep time divided by the total time in bed (that is, the number of minutes from the beginning of the Polysomnography recording to the end of the recording).
Effect of JNJ-54175446 Versus Placebo on Snaith-Hamilton Pleasure Scale [SHAPS]) | Baseline, Day 3, 4, 5 and 10: 2 to 8 hours postdose
  The SHAPS is a short, 14-item instrument to measure anhedonia, which has been shown to be valid and reliable in normal and clinical samples. Each of the 14 items has a set of four response categories: Definitely Agree (= 1), Agree (= 2), Disagree (= 3), and Definitely Disagree (= 4). A higher total score indicates higher levels of state anhedonia.
Effect of JNJ-54175446 Versus Placebo on Profile of Mood States brief form (POMS) | Baseline, Day 3, 10: 2 to 8 hours postdose, Day 4, 5: 2 to 8 and 19 hours postdose
  The POMS measures individuals' mood states. The POMS consists of 30 positive and negative mood descriptors. Participants are asked to rate, on a 5-point scale from 0 (not at all) to 4 (extremely), the extent to which they experience each mood state during at a specific moment.
Effect of JNJ-54175446 Versus Placebo on Emotional Faces Recognition Test | Baseline, Day 4 and 10: 2 to 8 hours postdose
  Evaluation of positive and negative effect using emotional faces recognition test. The participant is seated at a computer screen and instructed to remember 42 images shown during a training session. Subject then identifies those images during a testing session in which the 42 probe images are interspersed among 42 additional foil images. Implicit recognition is detected by EEG.
Effect of JNJ-54175446 Versus Placebo on Soluble Biomarkers (Inclusive Ex-vivo Lipopolysaccharide [LPS]/Benzoylated(Bz) Adenosine Triphosphate [ATP]-Induced IL-1 Beta Release) | Day 1 and 4: Predose, 2, 8 hours postdose, Day 10: Predose
Effect of JNJ-54175446 Versus Placebo on Central Pharmacodynamic (PD) by Motor Learning by Adaptive Tracking Test | Baseline, Day 10: Predose, 1, 2, 4 and 6 hour post dose
  Performance will be scored after a fixed period of 3.5 minutes and reflected visuo motor control and vigilance. The average performance scores will be used in the analysis.
Effect of JNJ-54175446 Versus Placebo on Sustained Attention by the Three Choice Vigilance Task (3CVT) With EEG | Baseline, Day 3, 4, 5 and 10: 2 to 8 hours postdose
  An implicit image recognition (IR) task combined with emotional elicitation evaluates attention, encoding and image recognition memory during implicit emotion elicitation.
Maximum Observed Plasma Concentration (Cmax) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  The Cmax is the maximum observed plasma concentration.
Minimum Observed Plasma Concentration (Cmin) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  Minimum observed plasma concentration during dosing interval (tau).
Trough Plasma Concentration (Ctrough) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  The observed plasma concentration just prior to the beginning or at the end of a dosing interval of any dose other than the first dose.
Average Plasma Concentration at Steady State (Cavg) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  Average plasma concentration at steady state over the dosing interval.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
Area Under the Plasma ConcentrationTime Curve During a Dosing Interval (tau) [AUCtau] of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
Area Under the Plasma ConcentrationTime Curve From Time Zero to Time 't' (AUC[0t]) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
Apparent Elimination HalfLife (t1/2) of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  Apparent elimination half-life associated with the terminal slope (Lambda[z]) of the semilogarithmic drug concentration time curve, after multiple-dose administration only.
Ratio of the Maximum Plasma Concentration (Peak) to Trough Observed Concentration of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  The ratio of the maximum plasma concentration (Peak) to trough observed concentration.
Accumulation Ratio Based on AUC of JNJ-54175446 | Day 1: Predose, 1, 2, 4, 8, 10 hour postdose; Day 2 and 3: Predose; Day 4: Predose, 2, 4, 8 hour postdose; Day 5 and 7: Predose; Day 10: Predose, 1, 2, 4, 8, 10, 24, 48 hour postdose; Day 17
  Accumulation ratio based on AUC, determined after multiple-dose administration and calculated as AUCtau on Day 1 divided by AUCtau on Day 10.
Effect of JNJ-54175446 Versus Placebo on a Reward Test | Baseline, Day 3, 4, 5 and 10: 2 to 8 hours postdose
  The reward task was a probabilistic instrumental learning task involving monetary wins or losses. In order to maximize payoffs, participants should use the outcome feedback to gradually learn the symbol-outcome associations by trial and error over time, such that they consistently choose the symbol with the high-probability win and avoid the symbol with the high-probability loss. Outcome measures included overall total, total won and lost, choice frequency, percentage of choices identical to the preceding one (percentage consistency), reaction time and re-reaction time.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Germany (3):
  - Berlin
  - Hamburg
  - Schwerin
- Leiden, Netherlands